CLINICAL TRIAL: NCT05795764
Title: Moderators of the Effectiveness of Crisis Response Planning (CRP) for Military Personnel
Brief Title: Crisis Response Planning for Military Personnel
Acronym: ASPIS/CRP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: United States Naval Medical Center, San Diego (U.S. Federal Agency)
Collaborators: Naval Health Research Center (U.S. Federal Agency); Ohio State University (Other)
Responsible Party: Principal Investigator, Kristen Walter, Principal Investigator, United States Naval Medical Center, San Diego
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NMCSD.2022.0058
Record Dates: First submitted 2023-03-10; First posted 2023-04-03 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Suicidal; Suicide Threat; Suicidal Ideation
MeSH Terms: conditions — Suicidal Ideation | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Crisis Response Planning (Experimental): CRP is a brief psychotherapeutic intervention that can be provided to patients at risk of suicidal behavior. When using the intervention, a provider works with the patient (1) to conduct a narrative assessment of the events preceding suicidal thoughts or behavior, and (2) to develop a personalized plan for identifying and managing distress that could escalate to a suicide attempt. The CRP, which is typically handwritten by the patient on an index card, includes personal warning signs of distress, emotion regulation strategies, reasons for living, and contact information for friends/family as well as professional (psychological/medical) and emergency resources.
  Interventions: Behavioral: Crisis Response Planning
- Treatment as Usual (Active Comparator): Existing clinical practices in the emergency department include the following elements recommended by the VA/DoD Clinical Practice Guidelines: (1) all patients are screened for suicidal ideation at every visit; (2) for those with positive screens, a suicide risk assessment interview is conducted by a mental health professional; (3) a safety planning form with means restriction (such as the Stanley-Brown; Stanley & Brown, 2012) is completed; and (4) patients are referred for follow-up mental health treatment as needed. Other elements of TAU could include behavioral and psychotropic interventions, referrals to specialty mental healthcare, and admission for psychiatric inpatient care.
  Interventions: Behavioral: Treatment as Usual

INTERVENTIONS:
Behavioral: Crisis Response Planning — Crisis Response Planning (CRP) is a brief psychotherapeutic intervention.
  Other Names: CRP
  Arms: Crisis Response Planning
Behavioral: Treatment as Usual — Standard care provided for patients at risk for suicide
  Arms: Treatment as Usual

SUMMARY:
The study is a randomized trial comparing outcomes of active duty service members who present to the emergency department at risk for suicide and receive care from providers trained in crisis response planning versus those providing treatment as usual.

ELIGIBILITY:
Inclusion Criteria:

* Active duty service members
* >18 years old
* Present to the emergency department at NMCSD with a primary concern related to suicidal ideation, plan, intention, or attempt, or are assessed as being at elevated risk of suicidal behavior
* Able to understand and speak English
* Able to provide consent

Exclusion Criteria:

* Unable to provide informed consent due to impaired mental status (e.g., acute intoxication, psychosis, mania, altered consciousness)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2023-06-21 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Self-Injurious Thoughts and Behaviors Interview (SITBI-R) | Through study completion, an average of 1 year
  Assessment of suicide attempts
Scale for Suicidal Ideation (SSI) | Through study completion, an average of 1 year
  Assessment of suicidal ideation; 19 items rated on a scale 0-2, higher scores indicate greater suicidal ideation severity

CONTACTS AND LOCATIONS:
Overall Officials: Kristen H Walter, PhD, Principal Investigator — Naval Health Research Center
Locations (1):
- Naval Medical Center San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: Yes
This study is one of five studies part of a consortium, referred to as ASPIS. All de-identified demographic and clinical data collected as part of the ASPIS projects will be available as raw individual-level data for sharing with external researchers working at an institution with a Federalwide Assurance (FWA) for the Protection of Human Subjects. ASPIS data will therefore be available for secondary analytic purposes. Names and institutions of persons either given or denied access to data will be tracked by our Administrative Core and will be available upon request from the sponsor. ASPIS data will not be available for data sharing until after all ASPIS projects are complete and the primary outcomes for each project are published.
Supporting Information: Study Protocol, ICF

REFERENCES:
- [Derived] Walter KH, Khandekar PR, Kline AC, Miggantz EL, Otis NP, Glassman LH, Thomsen CJ, Brock G, Bryan CJ. Comparison of crisis response planning and treatment as usual for active duty service members at risk for suicide: Study protocol for a stepped-wedge cluster randomized trial in a military treatment facility. Contemp Clin Trials Commun. 2024 Dec 6;42:101407. doi: 10.1016/j.conctc.2024.101407. eCollection 2024 Dec. PMID 39735169